CLINICAL TRIAL: NCT03318315
Title: A Phase II Study in Healthy Adults (19-64 Years of Age) to Assess the Safety, Reactogenicity and Immunogenicity of Sequential or Simultaneous Intramuscular Administration of an AS03-adjuvanted A/H7N9 Inactivated Influenza Vaccine With Seasonal Influenza Vaccine
Brief Title: Co-Administration of AS03 Adjuvanted A/H7N9 IIV With IIV4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-0077; HHSN272201300022I
Record Dates: First submitted 2017-10-19; First posted 2017-10-23 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2018-02-14

CONDITIONS: Avian Influenza; Influenza; Influenza Immunisation
Keywords: AS03-adjuvanted Inactivated Influenza Vaccine; Co-Administered; Healthy Adults; Immunogenicity; Inactivated Seasonal Influenza Vaccine; Phase II; Safety
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): 3.75 mcg HA per 0.5 mL dose of H7N9 vaccine in PBS diluent + GSK AS03 adjuvant and 0.5 ml dose of IIV4 vaccine, both administered intramuscularly within 15 minutes on day 1, and 3.75 mcg HA per 0.5 mL dose of H7N9 vaccine in PBS diluent + GSK AS03 adjuvant intramuscularly on day 22, n=60
  Interventions: Drug: AS03; Biological: Inactivated influenza H7N9 vaccine; Biological: Influenza Virus Quadrivalent Inactivated Vaccine; Other: Phosphate Buffered Saline (PBS) diluent
- Group 2 (Experimental): 0.5 ml dose of IIV4 vaccine intramuscularly on day 1 and 3.75 mcg HA per 0.5 ml dose of H7N9 vaccine in PBS diluent + GSK AS03 adjuvant intramuscularly on day 22 and day 43, n=60
  Interventions: Drug: AS03; Biological: Inactivated influenza H7N9 vaccine; Biological: Influenza Virus Quadrivalent Inactivated Vaccine; Other: Phosphate Buffered Saline (PBS) diluent
- Group 3 (Active Comparator): 0.5 ml dose of IIV4 vaccine intramuscularly on day 1, n=30
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine

INTERVENTIONS:
Drug: AS03 — AS03 oil-in-water emulsion adjuvant.
  Arms: Group 1; Group 2
Biological: Inactivated influenza H7N9 vaccine — Monovalent 2017 H7N9 inactivated influenza vaccine
  Arms: Group 1; Group 2
Biological: Influenza Virus Quadrivalent Inactivated Vaccine — A seasonal quadrivalent inactivated influenza vaccine (IIV4), prepared from influenza viruses propagated in embryonated chicken eggs, protecting against 2 influenza A subtypes (H1N1 and H3N2) and 2 influenza B subtypes (B Yamata lineage and B Victoria lineage).
Other: Phosphate Buffered Saline (PBS) diluent — Diluent for Adjuvanted 2017 Monovalent Inactivated Influenza A/H7N9 vaccine (2017 H7N9IIV)
  Arms: Group 1; Group 2

SUMMARY:
This is a randomized, un-blinded, Phase II study in males and non-pregnant females, who are in good health, 19 to 64 years of age. This study is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic AS03 (GSK) adjuvanted 2017 monovalent inactivated influenza A/H7N9 vaccine, when two doses are administered 21 days apart either sequentially or simultaneously (within 15 minutes) with licensed seasonal influenza vaccine. Subjects will be randomized into one of three treatment groups. The study will enroll approximately 150 individuals who have no history of influenza A/H7N9 infection or prior receipt of an influenza virus H7 subtype vaccine. Study duration is approximately 16 months with subject participation duration of approximately 13 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity following sequential or simultaneous IM administration of 2 doses of AS03-adjuvanted 2017 H7N9 IIV and one dose of seasonal influenza vaccine (IIV4); 2) to assess the serum HAI and Neut antibody responses against A/H7N9 at approximately 21 days following receipt of two doses of AS03-adjuvanted 2017 H7N9 IIV administered IM approximately 21 days apart; 3) to assess the serum HAI and Neut antibody responses against the seasonal influenza strains at approximately 21 days following receipt of IIV4.

DETAILED DESCRIPTION:
This is a randomized, un-blinded, Phase II study in males and non-pregnant females, who are in good health, 19 to 64 years of age. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic AS03 (GSK) adjuvanted 2017 monovalent inactivated influenza A/H7N9 vaccine (2017 H7N9 IIV) manufactured by Sanofi Pasteur (3.75 mcg of HA per dose with Phosphate Buffered Saline (PBS) diluent), when two doses are administered 21 days apart either sequentially or simultaneously (within 15 minutes) with licensed seasonal influenza vaccine. Subjects will be randomized into one of three treatment groups. Group 1 will receive two doses of AS03-adjuvanted 2017 H7N9 IIV, each dose administered IM approximately 21 days apart, and one dose of licensed seasonal IIV4 will be administered IM simultaneously (within 15 minutes) with the first dose of AS03 adjuvanted 2017 H7N9 IIV. Group 2 will receive one dose of IIV4 approximately 21 days prior to the IM administration of two doses of AS03-adjuvanted 2017 H7N9 IIV; each dose of AS03-adjuvanted 2017 H7N9 IIV will be given approximately 21 days apart. Group 3 will receive one dose IM of IIV4 as an un-blinded comparator. The study will enroll approximately 150 individuals who have no history of influenza A/H7N9 infection or prior receipt of an influenza virus H7 subtype vaccine. Study duration is approximately 16 months with subject participation duration of approximately 13 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity following sequential or simultaneous IM administration of 2 doses of AS03-adjuvanted 2017 H7N9 IIV and one dose of seasonal influenza vaccine (IIV4); 2) to assess the serum HAI and Neut antibody responses against A/H7N9 at approximately 21 days following receipt of two doses of AS03-adjuvanted 2017 H7N9 IIV administered IM approximately 21 days apart; 3) to assess the serum HAI and Neut antibody responses against the seasonal influenza strains at approximately 21 days following receipt of IIV4. The secondary objectives are: 1) to assess unsolicited non-SAEs following sequential or simultaneous IM administration of AS03-adjuvanted 2017 H7N9 IIV and seasonal influenza vaccine (IIV4); 2) to assess MAAEs, including NOCMCs and PIMMCs, following sequential or simultaneous IM administration of AS03-adjuvanted 2017 H7N9 IIV and IIV4; 3) to assess the HAI and Neut antibody responses at 21 days following receipt of 1 dose of AS03-adjuvanted 2017 H7N9 IIV.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 19 -64 years of age, inclusive.
4. Are in good health. - As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, Emergency Room (ER), or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.0°F.
6. Pulse is 47 to 100 beats per minute (bpm), inclusive.
7. Systolic blood pressure is 85 to 150 mmHg, inclusive (subjects <65 years of age), 85 to 160 mmHg, inclusive (subjects = / > 65 years of age).
8. Diastolic blood pressure is 55 to 95 mmHg, inclusive.
9. ESR is less than 30 mm per hour.
10. Women of childbearing potential must use an acceptable contraception method from 30 days before first study vaccination until 60 days after last study vaccination.

    - Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

    -- Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
11. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination.

   - An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation.

   - Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
7. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
8. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
9. Have a personal or family history of narcolepsy.
10. Have a history of Guillian-Barre Syndrome (GBS).
11. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
12. Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).
13. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
14. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
15. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
16. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
17. Have taken high-dose inhaled corticosteroids within 30 days prior to each study vaccination.

    - High-dose defined per age as using inhaled high dose per reference chart https://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines/quick-reference-html#estimated-comparative-daily-doses
18. Received a licensed live vaccine within 30 days prior to the first study vaccination, or plan to receive a licensed live vaccine within 30 days before or after each study vaccination.
19. Received or plan to receive a licensed, inactivated, vaccine (excluding all flu vaccines) within 14 days before or after each study vaccination.
20. Received or plan to receive the 2017-2018 inactivated seasonal flu vaccine prior to or during the clinical trial and for the remainder of the 2017-2018 season.
21. Received Ig or other blood products (with exception of Rho D Ig) within 90 days prior to each study vaccination.
22. Received an experimental agent within 30 days prior to the first study vaccination, or expect to receive an experimental agent during the 13-month trial-reporting period.

    - Including vaccine, drug, biologic, device, blood product, or medication.

    -- Other than from participation in this trial.
23. Are participating or plan to participate in another clinical trial with an interventional agent that will be received during the 13-month trial-reporting period.

    - Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
24. Received or plan to receive an influenza A/H7 vaccine or have a history of influenza A/H7 subtype infection.

    - And assigned to a group receiving influenza A/H7 vaccine.
25. Have traveled to mainland China and had substantial direct contact with live or freshly slaughtered poultry or pigeons within the past five years.

    - Substantial contact is defined as visited a poultry farm and/or a live poultry market.
26. Occupational exposure to or substantial direct physical contact with birds in the past year and through the 21 days after the last study vaccination.

    - Exposure to free range chickens in the yard is exclusionary. Casual contact with birds at petting zoos or county or state fairs, or having pet birds does not exclude subjects from study participation.
27. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
28. Plan to travel outside the US (continental US, Hawaii, and Alaska) from enrollment through 21 days after the last study vaccination.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham School of Medicine - Alabama Vaccine Research Clinic, Birmingham, Alabama
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University Medical Center - Infectious Diseases, Nashville, Tennessee

REFERENCES:
- [Derived] El Sahly HM, Anderson EJ, Jackson LA, Neuzil KM, Atmar RL, Bernstein DI, Chen WH, Creech CB, Frey SE, Goepfert P, Meier J, Phadke V, Rouphael N, Rupp R, Stapleton JT, Spearman P, Walter EB, Winokur PL, Yildirim I, Williams TL, Oshinsky J, Coughlan L, Nijhuis H, Pasetti MF, Krammer F, Stadlbauer D, Nachbagauer R, Tsong R, Wegel A, Roberts PC. Anti-neuraminidase and anti-hemagglutinin stalk responses to different influenza a(H7N9) vaccine regimens. Vaccine. 2025 Feb 15;47:126689. doi: 10.1016/j.vaccine.2024.126689. Epub 2025 Jan 4. PMID 39756216
- [Derived] Ortiz JR, Spearman PW, Goepfert PA, Cross K, Buddy Creech C, Chen WH, Parker S, Overton ET, Dickey M, Logan HL, Wegel A, Neuzil KM. Safety and immunogenicity of monovalent H7N9 influenza vaccine with AS03 adjuvant given sequentially or simultaneously with a seasonal influenza vaccine: A randomized clinical trial. Vaccine. 2022 May 20;40(23):3253-3262. doi: 10.1016/j.vaccine.2022.03.055. Epub 2022 Apr 22. PMID 35465983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult participants 19-64 years of age were recruited from the communities surrounding each clinical site, and were enrolled between 20FEB2018 and 29JUN2018.
Groups:
- Group 1 Simultaneous Administration: 3.75 mcg HA per 0.5 mL dose of Monovalent 2017 H7N9 inactivated influenza vaccine in Phosphate Buffered Saline (PBS) diluent + GSK AS03 adjuvant and 0.5 ml dose of seasonal quadrivalent inactivated influenza vaccine (IIV4), both administered intramuscularly within 15 minutes on Day 1, and 3.75 mcg HA per 0.5 mL dose of H7N9 vaccine in PBS diluent + GSK AS03 adjuvant intramuscularly on Day 22
- Group 2 Sequential Administration: 0.5 ml dose of IIV4 vaccine intramuscularly on day 1 and 3.75 mcg HA per 0.5 ml dose of H7N9 vaccine in PBS diluent + GSK AS03 adjuvant intramuscularly on Day 22 and Day 43
- Group 3 IIV4 Only: 0.5 ml dose of IIV4 vaccine intramuscularly on Day 1, n=30
Period: Overall Study
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Started | 62 | 53 | 34
Received First Vaccination | 62 | 53 | 34
Received Second Vaccination | 59 | 48 | 0
Received Third Vaccination | 0 | 46 | 0
Completed | 58 | 50 | 30
Not Completed | 4 | 3 | 4
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all randomized participants.
Groups:
- Group 1 Simultaneous Administration: 3.75 mcg HA of H7N9 IIV in PBS + GSK AS03 adjuvant and 0.5 ml IIV4, both administered IM within 15 minutes on Day 1, and 3.75 mcg HA of H7N9 vaccine in PBS + GSK AS03 adjuvant IM on Day 22
- Group 2 Sequential Administration: 0.5 ml dose of IIV4 vaccine IM on day 1 and 3.75 mcg HA of H7N9 vaccine in PBS + GSK AS03 adjuvant IM on Day 22 and Day 43
- Group 3 IIV4 Only: 0.5 ml dose of IIV4 vaccine IM on Day 1, n=30
- Total: Total of all reporting groups
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only | Total
Number analyzed (Participants) | 62 | 53 | 34 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 62 | 53 | 34 | 149
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (13.1) | 38.1 (11.5) | 35.7 (10.6) | 38.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 13 | 65
  Male | 36 | 27 | 21 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 52 | 31 | 143
  Not Hispanic or Latino | 2 | 1 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 36 | 29 | 17 | 82
  White | 22 | 17 | 14 | 53
  More than one race | 1 | 4 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 53 | 34 | 149

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies Against the 2017 H7N9 Inactivated Influenza Vaccine (IIV) Strain After Second H7N9 Vaccination
Description: Blood was collected for HAI assay at conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days after the second dose of H7N9, which is Day 43 for Group 1 and Day 64 for Group 2.
Time Frame: 21 days after second dose of H7N9
Population: Participants included in the modified intent-to-treat (mITT) population are those who received the first study dose have immunogenicity results at baseline and at least one timepoint post baseline. If baseline results are unavailable for an assay at baseline, the participant is not included in mITT analysis at any timepoint for that assay only.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 47
titer | 36.8 [27.7 to 48.8] | 22.7 [16.9 to 30.6]

2. Primary Outcome: GMTs of Serum HAI Antibodies Against Each of the 2017 IIV4 Strains
Description: Blood was collected for HAI assay at conducted with the IIV4 vaccine viruses as the antigens. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results.
Time Frame: Day 22
Population: Participants included in the mITT population are those who received the first study dose have immunogenicity results at baseline and at least one timepoint post baseline. If baseline results are unavailable for an assay at baseline, the participant is not included in mITT analysis at any timepoint for that assay only.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 55 | 52 | 29
titer
  A/Michigan/45/2015 x-275 (H1N1) | 547.7 [431.0 to 696.1] | 503.6 [360.6 to 703.1] | 480.4 [290.1 to 795.7]
  A/Hong Kong/4801/2014 X-263B (H3N2) | 284.0 [201.6 to 400.0] | 289.8 [202.5 to 414.7] | 462.6 [314.6 to 680.2]
  B/Phuket/3073/2013 (B Yamagata lineage) | 20.8 [15.2 to 28.4] | 23.05 [17.3 to 31.9] | 44.4 [29.7 to 66.3]
  B/Brisbane/60/2008 (B Victoria lineage) | 46.1 [33.6 to 63.2] | 61.8 [46.0 to 82.9] | 64.1 [44.3 to 92.7]

3. Primary Outcome: GMTs of Serum Neutralizing Antibodies Against Each of the 2017 IIV4 Strains
Description: Blood was collected for the serum neutralizing antibody assay conducted with the IIV4 vaccine viruses as the antigens. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results.
Time Frame: Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 54 | 52 | 29
titer
  A/Michigan/45/2015 x-275 (H1N1) | 230.4 [169.2 to 313.6] | 186.0 [123.0 to 281.1] | 227.6 [133.9 to 386.9]
  A/Hong Kong/4801/2014 X-263B (H3N2) | 481.3 [343.7 to 674.0] | 518.4 [358.1 to 750.5] | 788.9 [584.0 to 1065.6]
  B/Phuket/3073/2013 (B Yamagata lineage) | 237.9 [176.8 to 320.0] | 251.5 [193.9 to 326.2] | 452.5 [327.7 to 625.0]
  B/Brisbane/60/2008 (B Victoria lineage) | 118.9 [90.5 to 156.3] | 157.4 [117.9 to 210.2] | 202.0 [145.0 to 281.4]

4. Primary Outcome: GMTs of Serum Neutralizing Antibodies Against the 2017 H7N9 IIV Strain After the Second H7N9 Vaccination
Description: Blood was collected for the serum neutralizing antibody assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days after second dose of H7N9, which is Day 43 for Group 1 and Day 64 for Group 2.
Time Frame: 21 days after second dose of H7N9
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 47
titer | 88.4 [63.2 to 123.9] | 50.5 [37.4 to 68.0]

5. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All events are included regardless of relationship to the study product.
Time Frame: Day 1 up to Day 408
Population: The safety population includes all subjects receiving study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants | 0 | 1 | 0

6. Primary Outcome: Number of Participants Assessed With Clinical Safety Laboratory AEs After First Vaccination
Description: Laboratory parameters include alanine aminotransferase (ALT), bilirubin, creatinine, hemoglobin, platelets and white blood cells (WBC). Thresholds for adverse events were considered as ALT 44 IU/L or greater (female) or 61 IU/L or greater (male); bilirubin 1.30 mg/dL or greater; creatinine 1.1 mg/dL or greater (female) or 1.4 mg/dL or greater (male); hemoglobin 11.4 g/dL or lower (female) or 12.4 g/dL or lower (male); platelets 139 x10^3/µL or below or 416 x10^3/µL or greater; or WBC or 3.9 x10^3/µL or lower or 10.6 x10^3/µL or higher.
Time Frame: Day 8
Population: The safety population includes all subject receiving study product with data at the time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants
  ALT | 3 | 1 | 0
  bilirubin | 1 | 0 | 0
  creatinine | 3 | 0 | 0
  hemoglobin | 4 | 6 | 3
  platelets | 1 | 1 | 0
  WBC | 5 | 4 | 2

7. Primary Outcome: Number of Participants Assessed With Clinical Safety Laboratory AEs After Second Vaccination
Description: as for outcome 6
Time Frame: Day 29
Population: The safety population includes all subject receiving study product with data at the time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 47
Participants
  ALT | 5 | 0
  bilirubin | 1 | 1
  creatinine | 1 | 0
  hemoglobin | 2 | 4
  platelets | 3 | 0
  WBC | 3 | 6

8. Primary Outcome: Number of Participants Assessed With Clinical Safety Laboratory AEs After Third Vaccination
Description: as for outcome 6
Time Frame: Day 50
Population: The safety population includes all subject receiving study product with data at the time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 Sequential Administration
Number analyzed (Participants) | 44
Participants
  ALT | 0
  bilirubin | 0
  creatinine | 1
  hemoglobin | 4
  platelets | 1
  WBC | 5

9. Primary Outcome: Number of Participants Reporting Solicited Injection Site AEs After First Vaccination
Description: Injection site AEs solicited on a memory aid provided to participants included . Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days following vaccination Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (measurement grade)
Time Frame: Day 1 up to day 8
Population: The safety population includes all subject receiving study product with data reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants
  Pain | 44 | 18 | 14
  Tenderness | 44 | 30 | 17
  Itching/Pruritus | 5 | 2 | 2
  Ecchymosis/Bruising (functional grade) | 4 | 2 | 1
  Ecchymosis/Bruising (measured) | 4 | 2 | 1
  Erythema/Redness (functional grade) | 15 | 5 | 4
  Erythema/Redness (measured) | 14 | 5 | 4
  Induration/Swelling (functional grade) | 13 | 5 | 0
  Induration/Swelling (measured) | 11 | 5 | 0

10. Primary Outcome: Number of Participants Reporting Solicited Injection Site AEs After Second Vaccination
Description: as for outcome 9
Time Frame: Day 22 up to day 29
Population: The safety population includes all subject receiving study product with data reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 48
Participants
  Pain | 24 | 24
  Tenderness | 32 | 32
  Itching/Pruritus | 4 | 3
  Ecchymosis/Bruising (functional grade) | 5 | 2
  Ecchymosis/Bruising (measured) | 5 | 2
  Erythema/Redness (functional grade) | 13 | 7
  Erythema/Redness (measured) | 12 | 7
  Induration/Swelling (functional grade) | 13 | 9
  Induration/Swelling (measured) | 12 | 9

11. Primary Outcome: Number of Participants Reporting Solicited Injection Site AEs After Third Vaccination
Description: as for outcome 9
Time Frame: Day 43 up to day 50
Population: The safety population includes all subject receiving study product with data reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 Sequential Administration
Number analyzed (Participants) | 46
Participants
  Pain | 17
  Tenderness | 30
  Itching/Pruritus | 2
  Ecchymosis/Bruising (functional grade) | 2
  Ecchymosis/Bruising (measured) | 2
  Erythema/Redness (functional grade) | 4
  Erythema/Redness (measured) | 4
  Induration/Swelling (functional grade) | 5
  Induration/Swelling (measured) | 5

12. Primary Outcome: Occurrence of Study Vaccine-related SAEs
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. Events are included if deemed by the investigator to be related to the study product.
Time Frame: Day 1 up to day 408
Population: The safety population includes all subjects receiving study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants | 0 | 0 | 0

13. Primary Outcome: Number of Participants Reporting Solicited Systemic AEs After First Vaccination
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days following vaccination.
Time Frame: Day 1 up to day 8
Population: The safety population includes all participants receiving the dose and for whom solicited data were reported
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants
  Elevated Oral Temperature | 1 | 0 | 2
  Feverishness | 13 | 0 | 3
  Fatigue | 25 | 11 | 7
  Malaise | 19 | 6 | 8
  Myalgia | 28 | 7 | 9
  Arthralgia | 8 | 4 | 4
  Headache | 17 | 7 | 8
  Nausea | 2 | 1 | 5

14. Primary Outcome: Number of Participating Reporting Solicited Systemic AEs After Second Vaccination
Description: as for outcome 13
Time Frame: Day 22 up to day 29
Population: The safety population includes all participants receiving the dose and for whom solicited data were reported
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 48
Participants
  Elevated Oral Temperature | 0 | 1
  Feverishness | 8 | 7
  Fatigue | 17 | 14
  Malaise | 13 | 9
  Myalgia | 19 | 8
  Arthralgia | 9 | 5
  Headache | 13 | 8
  Nausea | 6 | 6

15. Primary Outcome: Number of Participants Reporting Solicited Systemic AEs After Third Vaccination
Description: as for outcome 13
Time Frame: Day 43 up to day 50
Population: The safety population includes all participants receiving the dose and for whom solicited data were reported
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 Sequential Administration
Number analyzed (Participants) | 46
Participants
  Elevated Oral Temperature | 0
  Feverishness | 2
  Fatigue | 10
  Malaise | 5
  Myalgia | 11
  Arthralgia | 4
  Headache | 4
  Nausea | 3

16. Primary Outcome: Percentage of Participants Achieving HAI Seroconversion Against 2017 H7N9 Study Vaccine After Second H7N9 Vaccination
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer = / >1:40 or pre-vaccination titer 1:10 or greater and min. 4-fold rise in post-vaccination antibody titer. 21 days after second dose of H7N9 is Day 22 for Group 1 and Day 43 for Group 2.
Time Frame: 21 days after second dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 47
percentage of participants | 51 [37 to 64] | 38 [25 to 54]

17. Primary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion Against 2017 H7N9 Study Vaccine After Second H7N9 Vaccination
Description: Blood was collected for the serum neutralizing antibody assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as neutralizing antibody pre-vaccination titer <1:10 and post-vaccination titer 1:40 or greater, or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second dose of H7N9 is Day 22 for Group 1 and Day 43 for Group 2.
Time Frame: 21 days after second dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 47
percentage of participants | 82 [70 to 91] | 74 [60 to 86]

18. Primary Outcome: Percentage of Participants Achieving HAI Seroconversion Against Each of the Study IIV4 Strains
Description: Blood was collected for the HAI assay conducted with the IIV4 vaccine viruses as the antigens. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer = / >1:40 or pre-vaccination titer 1:10 or greater and min. 4-fold rise in post-vaccination antibody titer.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 59 | 53 | 29
percentage of participants
  A/Michigan/45/2015 x-275 (H1N1) | 53 [39 to 66] | 58 [44 to 72] | 55 [36 to 74]
  A/Hong Kong/4801/2014 X-263B (H3N2) | 49 [36 to 63] | 55 [40 to 68] | 72 [53 to 87]
  B/Phuket/3073/2013 (B Yamagata lineage) | 19 [10 to 31] | 13 [5 to 25] | 41 [24 to 61]
  B/Brisbane/60/2008 (B Victoria lineage) | 29 [18 to 42] | 47 [33 to 61] | 48 [29 to 67]

19. Primary Outcome: Percentage of Participants With HAI Antibody Titer of 1:40 or Greater Against Each of the Study IIV4 Strains
Description: Blood was collected for the HAI assay conducted with the IIV4 vaccine viruses as the antigens. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 59 | 53 | 29
percentage of participants
  A/Michigan/45/2015 x-275 (H1N1) | 100 [94 to 100] | 96 [87 to 100] | 93 [77 to 99]
  A/Hong Kong/4801/2014 X-263B (H3N2) | 93 [84 to 98] | 94 [84 to 99] | 100 [88 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) | 25 [15 to 38] | 30 [18 to 44] | 62 [42 to 79]
  B/Brisbane/60/2008 (B Victoria lineage) | 54 [41 to 67] | 72 [58 to 83] | 76 [56 to 90]

20. Primary Outcome: Percentage of Participants With HAI Antibody Titer of 1:40 or Greater Against the Influenza 2017 H7N9 Study Vaccine Strain After Second H7N9 Vaccination
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. 21 days after second dose of H7N9 is Day 43 for Group 1 and Day 64 for Group 2
Time Frame: 21 days after second dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 47
percentage of participants | 51 [37 to 64] | 38 [25 to 54]

21. Primary Outcome: Percentage of Participants With Neutralizing Antibody Titer of 1:40 or Greater Against Each of the Study IIV4 Strains
Description: Blood was collected for the serum neutralizing antibody assay conducted with the IIV4 vaccine viruses as the antigens. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 58 | 53 | 29
percentage of participants
  A/Michigan/45/2015 x-275 (H1N1) | 98 [91 to 100] | 85 [72 to 93] | 93 [77 to 99]
  A/Hong Kong/4801/2014 X-263B (H3N2) | 93 [84 to 98] | 94 [84 to 99] | 100 [88 to 100]
  B/Phuket/3073/2013 (B Yamagata lineage) | 95 [86 to 99] | 100 [93 to 100] | 100 [88 to 100]
  B/Brisbane/60/2008 (B Victoria lineage) | 90 [79 to 96] | 96 [87 to 100] | 100 [88 to 100]

22. Primary Outcome: Percentage of Participants With Neutralizing Antibody Titer of 1:40 or Greater Against the Influenza 2017 H7N9 Study Vaccine Strain After Second H7N9 Vaccination
Description: Blood was collected for the serum neutralizing antibody assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. 21 days after second dose of H7N9 is Day 43 for Group 1 and Day 64 for Group 2
Time Frame: 21 days after second dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 47
percentage of participants | 84 [72 to 93] | 74 [60 to 86]

23. Secondary Outcome: GMTs of Serum HAI Antibodies Against the Influenza 2017 H7N9 Vaccine Virus at Baseline
Description: Blood was collected for HAI assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results.
Time Frame: Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 53
titer | 5.7 [5.5 to 6.0] | 5.7 [5.3 to 6.1]

24. Secondary Outcome: GMTs of Serum HAI Antibodies Against the Influenza 2017 H7N9 Vaccine Virus After First H7N9 Vaccination
Description: Blood was collected for HAI assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results. 21 days after first dose of H7N9 is Day 22 for Group 1 and Day 43 for Group 2.
Time Frame: 21 days after first dose of H7N9
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 50
titer | 9.9 [7.7 to 12.7] | 6.6 [5.9 to 7.4]

25. Secondary Outcome: GMTs of Serum Neutralizing Antibodies Against the Influenza 2017 H7N9 Vaccine Virus at Baseline
Description: Blood was collected for the serum neutralizing antibody assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results.
Time Frame: Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 60 | 53
titer | 5.9 [5.4 to 6.6] | 5.4 [5.1 to 5.7]

26. Secondary Outcome: GMTs of Serum Neutralizing Antibodies Against the Influenza 2017 H7N9 Vaccine Virus After First H7N9 Vaccination
Description: Blood was collected for serum neutralizing antibody assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results. 21 days after first dose of H7N9 is Day 22 for Group 1 and Day 43 for Group 2.
Time Frame: 21 days after first dose of H7N9
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 50
titer | 22.3 [16.2 to 30.8] | 18.4 [14.5 to 23.4]

27. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs After First Vaccination
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through approximately 21 days after each vaccination. Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Approximately 21 days after first vaccination
Population: The safety population includes all participants receiving the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants
  Any SOC | 18 | 11 | 4
  Blood And Lymphatic System Disorders | 0 | 1 | 0
  Eye Disorders | 0 | 1 | 0
  Gastrointestinal Disorders | 2 | 1 | 0
  General Disorders / Administration Site Conditions | 3 | 1 | 0
  Infections And Infestations | 8 | 2 | 3
  Injury, Poisoning And Procedural Complications | 0 | 1 | 0
  Investigations | 3 | 3 | 0
  Musculoskeletal And Connective Tissue Disorders | 1 | 0 | 1
  Nervous System Disorders | 3 | 1 | 0
  Psychiatric Disorders | 1 | 0 | 0
  Reproductive System And Breast Disorders | 1 | 0 | 0
  Respiratory, Thoracic And Mediastinal Disorders | 1 | 0 | 0
  Vascular Disorders | 0 | 1 | 0

28. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs After Second Vaccination
Description: as for outcome 27
Time Frame: Approximately 21 days after second vaccination
Population: The safety population includes all participants who received the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 48
Participants
  Any SOC | 12 | 6
  Gastrointestinal Disorders | 2 | 1
  General Disorders / Administration Site Conditions | 1 | 1
  Infections And Infestations | 5 | 2
  Injury, Poisoning And Procedural Complications | 1 | 0
  Investigations | 2 | 0
  Musculoskeletal And Connective Tissue Disorders | 2 | 0
  Nervous System Disorders | 1 | 1
  Psychiatric Disorders | 0 | 1

29. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs After Third Vaccination
Description: as for outcome 27
Time Frame: Approximately 21 days after third vaccination
Population: The safety population includes all participants who received the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 Sequential Administration
Number analyzed (Participants) | 46
Participants
  Any SOC | 4
  General Disorders / Administration Site Conditions | 1
  Investigations | 1
  Musculoskeletal And Connective Tissue Disorders | 1
  Nervous System Disorders | 1

30. Secondary Outcome: Number of Participants Reporting of Medically-Attended Adverse Events (MAAEs), Including New-Onset Chronic Medical Conditions (NOCMCs) and Potentially Immune-Mediated Medical Conditions (PIMMCs)
Description: Participants were queried at each visit for the occurrence of medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) throughout the duration of the study.
Time Frame: Day 1 up to day 408
Population: The safety population included all participants who received at least one dose of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants
  MAAE | 6 | 6 | 2
  NOCMC | 1 | 2 | 0
  PIMMC | 0 | 0 | 0

31. Secondary Outcome: Number of Participants Reporting Study Vaccine-related Unsolicited Non-serious AEs After First Vaccination
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through approximately 21 days after each vaccination. The site investigator determined vaccine related as "a reasonable possibility that the study product caused the AE. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the AE." Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Approximately 21 days after first vaccination
Population: The safety population includes all participants receiving the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
Number analyzed (Participants) | 62 | 53 | 34
Participants
  Any SOC | 7 | 2 | 0
  Gastrointestinal Disorders | 1 | 1 | 0
  General Disorders / Administration Site Conditions | 2 | 1 | 0
  Infections And Infestations | 1 | 0 | 0
  Investigations | 1 | 0 | 0
  Nervous System Disorders | 2 | 0 | 0
  Psychiatric Disorders | 1 | 0 | 0
  Respiratory, Thoracic And Mediastinal Disorders | 1 | 0 | 0

32. Secondary Outcome: Number of Participants Reporting Study Vaccine-related Unsolicited Non-serious AEs After Second Vaccination
Description: as for outcome 31
Time Frame: Approximately 21 days after second vaccination
Population: The safety population includes all participants receiving the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 48
Participants
  Any SOC | 3 | 3
  Gastrointestinal Disorders | 1 | 1
  General Disorders / Administration Site Conditions | 1 | 0
  Infections And Infestations | 0 | 1
  Musculoskeletal And Connective Tissue Disorders | 1 | 0
  Nervous System Disorders | 0 | 1

33. Secondary Outcome: Number of Participants Reporting Study Vaccine-related Unsolicited Non-serious AEs After Third Vaccination
Description: as for outcome 31
Time Frame: Approximately 21 days after third vaccination
Population: The safety population includes all participants receiving the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 Sequential Administration
Number analyzed (Participants) | 46
Participants
  Any SOC | 2
  Investigations | 1
  Nervous System Disorders | 1

34. Secondary Outcome: Percentage of Participants Achieving HAI Antibody Seroconversion Against the 2017 H7N9 Vaccine Strain After First H7N9 Vaccination
Description: Blood was collected for HAI assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer 1:40 or greater, or pre-vaccination titer 1:10 or greater and min. 4-fold rise in post-vaccination antibody titer. 21 days after first dose of H7N9 is Day 22 for Group 1 and Day 43 for Group 2.
Time Frame: 21 days after first dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 50
percentage of participants | 14 [6 to 26] | 2 [0 to 11]

35. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion Against the 2017 H7N9 Vaccine Strain After First H7N9 Vaccination
Description: Blood was collected for serum neutralizing antibody assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as a pre-vaccination titer <1:10 and post-vaccination titer 1:40 or greater, or pre-vaccination titer 1:10 or greater and min. 4-fold rise in post-vaccination antibody titer. 21 days after first dose of H7N9 is Day 22 for Group 1 and Day 43 for Group 2.
Time Frame: 21 days after first dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 50
percentage of participants | 34 [22 to 47] | 28 [16 to 42]

36. Secondary Outcome: Percentage of Participants Achieving Serum HAI Antibody Titers of 1:40 or Greater Against the Influenza 2017 H7N9 Vaccine Strain at Baseline
Description: Blood was collected for HAI assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 53
percentage of participants | 0 [0 to 6] | 0 [0 to 7]

37. Secondary Outcome: Percentage of Participants Achieving Serum HAI Antibody Titers of 1:40 or Greater Against the Influenza 2017 H7N9 Vaccine Strain After First H7N9 Vaccination
Description: Blood was collected for serum neutralizing antibody assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. 21 days after first H7N9 vaccination was Day 22 for Group 1 and Day 43 for Group 2
Time Frame: 21 days after first dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 57 | 50
percentage of participants | 14 [6 to 26] | 2 [0 to 11]

38. Secondary Outcome: Percentage of Participants Achieving Serum Neutralizing Antibody Titers of 1:40 or Greater Against the Influenza 2017 H7N9 Vaccine Strain at Baseline
Description: Blood was collected for serum neutralizing antibody assay at conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 60 | 53
percentage of participants | 2 [0 to 9] | 0 [0 to 7]

39. Secondary Outcome: Percentage of Participants Achieving Serum Neutralizing Antibody Titers of 1:40 or Greater Against the Influenza 2017 H7N9 Vaccine Strain After First H7N9 Vaccination
Description: as for outcome 37
Time Frame: 21 days after first dose of H7N9
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration
Number analyzed (Participants) | 59 | 50
percentage of participants | 34 [22 to 47] | 28 [16 to 42]

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 7 days after each vaccination, unsolicited non-serious AEs through 21 days after each vaccination, and SAEs through approximately 1 year after the last study vaccination.
Description: For events solicited on the Memory Aid in the 7 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 7-day period. Each 7-day period was considered a separate event.
Arm/Group | Group 1 Simultaneous Administration | Group 2 Sequential Administration | Group 3 IIV4 Only
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/53 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/62 | 1/53 | 0/34
Other Adverse Events (participants affected / at risk) | 57/62 | 48/53 | 25/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Simultaneous Administration (N=62) | Group 2 Sequential Administration (N=53) | Group 3 IIV4 Only (N=34)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Simultaneous Administration (N=62) | Group 2 Sequential Administration (N=53) | Group 3 IIV4 Only (N=34)
Nausea (Gastrointestinal disorders) | 7 (8) | 8 (10) | 5 (5)
Fatigue (General disorders) | 27 (42) | 23 (37) | 7 (7)
Feeling hot (General disorders) | 17 (21) | 9 (9) | 3 (3) — Solicited as "feverishness"
Injection site erythema (General disorders) | 20 (38) | 13 (16) | 4 (4)
Injection site haemorrhage (General disorders) | 8 (9) | 5 (6) | 1 (1)
Injection site induration (General disorders) | 19 (30) | 16 (19) | 0 (0)
Injection site pain (General disorders) | 45 (93) | 33 (59) | 14 (14) — Solicited as "Injection site pain"
Injection site pain (General disorders) | 48 (106) | 40 (92) | 17 (17) — Solicited as "Injection site tenderness"
Injection site pruritus (General disorders) | 9 (9) | 6 (7) | 2 (2)
Malaise (General disorders) | 24 (32) | 15 (20) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (11) | 1 (3) | 0 (0)
Blood creatinine increased (Investigations) | 4 (6) | 2 (3) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 1 (1) | 2 (2) — Defined as oral temperature of 100.4 degrees Fahrenheit or greater
Haemoglobin decreased (Investigations) | 4 (11) | 8 (24) | 3 (3)
Platelet count increased (Investigations) | 4 (8) | 2 (3) | 0 (0)
White blood cell count decreased (Investigations) | 4 (4) | 10 (24) | 0 (0)
White blood cell count increased (Investigations) | 9 (12) | 5 (9) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (17) | 9 (13) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 33 (47) | 17 (26) | 9 (9)
Headache (Nervous system disorders) | 27 (32) | 15 (20) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03318315/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03318315/SAP_001.pdf